CLINICAL TRIAL: NCT00235001
Title: A Multicenter, Open, Phase IV, 24-Hour Ambulatory Blood Pressure Monitoring Study of the Efficacy and Safety of Tarka in Patients With Arterial Hypertension
Brief Title: Russian Study of the Efficacy and Safety of Tarka in Patients With Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Peter Bacher, MD, PhD, Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RUSS-04-01
Record Dates: First submitted 2005-09-13; First posted 2005-10-10 (Estimated); Last update posted 2008-07-10 (Estimated); Status verified 2008-07

CONDITIONS: Hypertension
Keywords: Hypertension; Tarka
MeSH Terms: conditions — Hypertension | interventions — trandolapril; Verapamil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: trandolapril/verapamil

INTERVENTIONS:
Drug: trandolapril/verapamil — 180/2 mg QD
  Other Names: ABT-TARKA; Tarka

SUMMARY:
This study will investigate antihypertensive activity and safety profile of Tarka in Russian hypertension patients by ambulatory blood pressure measurement (ABPM)

ELIGIBILITY:
Inclusion Criteria:

* Hypertension

Exclusion Criteria:

* SBP > 180 mm Hg, DBP > 114 mm Hg
* Subject has a hypersensitivity to trandolapril or verapamil

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2004-06; Primary Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure from baseline/blood pressure control | Baseline to 3 months of Tx

SECONDARY OUTCOMES:
Absolute BP reduction from baseline, safety | Baseline to 3 months of Tx

CONTACTS AND LOCATIONS:
Overall Officials: Victor Gorin, MD, Study Director — Abbott
Locations (1):
- Global Medical Information-Abbott, North Chicago, Illinois, United States